CLINICAL TRIAL: NCT02297698
Title: Phase II Trial of Combination Immunotherapy With Nelipepimut-S + GM-CSF (NeuVax™) and Trastuzumab in High-risk HER2+ Breast Cancer Patients
Brief Title: Phase II Trial of Combination Immunotherapy With NeuVax and Trastuzumab in High-risk HER2+ Breast Cancer Patients
Acronym: HER3+
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Insight, LLC (Industry)
Collaborators: Genentech, Inc. (Industry); Sellas Life Sciences Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-0443
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer, NeuVax
MeSH Terms: conditions — Breast Neoplasms | interventions — HER2 peptide (369-377); Trastuzumab; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trastuzumab + NeuVax (Experimental): Patients randomized to this arm will receive vaccinations of nelipepimut-S (1000 μg) and GM-CSF (250 μg) (NeuVax vaccine) administered intradermally every three weeks for six total vaccinations, 30-120 minutes after completion of trastuzumab infusion. The first vaccination will be given with the third dose of maintenance trastuzumab administered as monotherapy optimally, but may be given with later maintenance doses of trastuzumab, provided there are at least six remaining doses of trastuzumbab to overlap with the PVS. Upon completion of the primary vaccination series (PVS), booster inoculations (same dose and route) will be administered every six months x 4. The first booster inoculation will occur 6 months ± 2 weeks after the completion of the PVS, with subsequent boosters timed every six months + 2 weeks. Boosters will therefore occur at the following time points after completion of the PVS: 6 months ± 2 weeks, 12 months ± 2 weeks, 18 months ± 2 weeks and 24 months ± 2 weeks.
  Interventions: Biological: NeuVax vaccine; Drug: Trastuzumab; Drug: GM-CSF
- Trastuzumab + GM-CSF (Active Comparator): Patients randomized to this arm will receive inoculations of GM-CSF (250 μg) administered in an identical manner to those receiving nelipepimut-S/GM-CSF (NeuVax). Patients will be blinded as to whether they are receiving nelipepimut-S/GM-CSF or GM-CSF alone. Upon completion of the primary vaccination series (PVS), booster inoculations (same dose and route) will be administered every six months x 4. The first booster inoculation will occur 6 months ± 2 weeks after the completion of the PVS, with subsequent boosters timed every six months + 2 weeks. Boosters will therefore occur at the following time points after completion of the PVS: 6 months ± 2 weeks, 12 months ± 2 weeks, 18 months ± 2 weeks and 24 months ± 2 weeks.
  Interventions: Drug: Trastuzumab; Drug: GM-CSF

INTERVENTIONS:
Biological: NeuVax vaccine — At the time of vaccine administration, a frozen solution of E75 acetate (1.5 mg/mL) is thawed and 1000mcg E75 peptide mixed thoroughly with 250mcg GM-CSF. This constitutes the NeuVax vaccine. Patients randomized to this arm will receive vaccinations of nelipepimut-S/GM-CSF administered intradermally every three weeks for six total vaccinations, 30-120 minutes after completion of trastuzumab infusion. The first vaccination will be given with the third dose of maintenance trastuzumab administered as monotherapy optimally, but may be given with later maintenance doses of trastuzumab, provided there are at least six remaining doses of trastuzumab to overlap with the primary vaccine series.
  Other Names: nelipepimut-S
  Arms: Trastuzumab + NeuVax
Drug: Trastuzumab — Herceptin will be administered to patients every three weeks as monotherapy for one year, to be given upon completion of standard of care chemotherapy/radiotherapy. The first trastuzumab infusion will be given no sooner than three weeks and no later than 12 weeks after completion of chemotherapy/radiotherapy. Trastuzumab will be dosed at the recommended initial loading dose of 8 mg/kg and at recommended maintenance doses of 6 mg/kg q3wk.
  Other Names: Herceptin
Drug: GM-CSF — For patients randomized to the GM-CSF alone arm, they will receive inoculations of GM-CSF (250mcg) administered intradermally every three weeks for six total vaccinations, 30-120 minutes after completion of trastuzumab infusion. The first injection will be given with the third dose of maintenance trastuzumab administered as monotherapy optimally, but may be given with later maintenance doses of trastuzumab, provided there are at least six remaining doses of trastuzumab to overlap with the primary vaccine series.
  Other Names: Leukine; Sargramostim

SUMMARY:
This will be a multi-center, prospective, randomized, single-blinded, placebo-controlled phase II trial of trastuzumab + nelipepimut-S/GM-CSF versus trastuzumab + GM-CSF alone. Our target study population is high-risk HER2-positive breast cancer patients. High-risk HER2-positive breast cancer patients are defined as:

Those with HER2-positive breast cancer, regardless of hormone receptor status, who receive neoadjuvant therapy with an approved regimen that includes trastuzumab and at least four cycles (12 weeks) of taxane-containing chemotherapy, and fail to achieve a pCR.

Those with HER2-positive breast cancer, regardless of hormone receptor status, who undergo surgery as a first intervention and are found to have ≥ 4 positive lymph nodes.

Those with HER2-positive, hormone receptor negative breast cancer who undergo surgery as a first intervention and are found to have 1-3 positive lymph nodes.

Disease-free subjects after standard of care multi-modality therapy will be screened and HLA-typed.

DETAILED DESCRIPTION:
In this study, the investigators intend to assess the ability of the combination of trastuzumab and the HER2 vaccine nelipepimut-S (administered with the immunoadjuvant GM-CSF) given in the adjuvant setting to prevent recurrences in patients with high-risk HER2-positive breast cancer. High-risk is defined as those patients that do not achieve a pCR after neoadjuvant therapy with an approved regimen that includes trastuzumab and at least four cycles (12 weeks) of taxane-containing chemotherapy or those who undergo upfront surgery and are found to have greater than or equal to four positive lymph nodes regardless of hormone receptor status or 1-3 positive lymph nodes and are hormone receptor negative.

Following surgery, patients will be screened and HLA-typed (consent #1). Nelipepimut-S is a CD8-eliciting peptide vaccine that is restricted to HLA-2+ or HLA-A3+ or HLA-A24+ or HLA-A26+ patients (approximately 80% of the US population). HLA-A2+/A3+/A24+/orA26+ patients who meet all other eligibility criteria will be randomized to receive trastuzumab + nelipepimut-S/GM-CSF or trastuzumab + GM-CSF alone (consent #2). The trastuzumab will be administered to all patients consistent with current standard of care. Patients randomized to the nelipepimut-S/GM-CSF arm will receive vaccinations of nelipepimut-S (1000 mcg) and GM-CSF (250 mcg) administered intradermally every three weeks for six total vaccinations, 30-120 minutes after completion of trastuzumab infusion. The first vaccination will be given with the third dose of maintenance trastuzumab administered as monotherapy optimally, but may be given with later maintenance doses of trastuzumab, provided there are at least six remaining doses of trastuzumab to overlap with the primary vaccine series. Patients randomized to the GM-CSF alone arm will receive inoculations of GM-CSF (250 mcg) administered in an identical manner to those receiving nelipepimut-S/GM-CSF. Patients will be blinded as to whether they are receiving nelipepimut-S/GM-CSF or GM-CSF alone.

Upon completion of the primary vaccination/inoculation series, booster inoculations (same dose and route) will be administered every six months x 4. The first booster inoculation will occur 6 months ± 2 weeks after the completion of the PVS, with subsequent boosters timed every six months + 2 weeks. Boosters will therefore occur at the following time points after completion of the PVS: 6 months ± 2 weeks, 12 months ± 2 weeks, 18 months ± 2 weeks, 24 months ± 2 weeks. Booster inoculations will occur for patients randomized to receive nelipepimut-S/GM-CSF as well as patients randomized to receive GM-CSF alone, and will consist of the same treatment drugs and dosing (i.e., nelipepimut-S/GM-CSF patients will be boosted with nelipepimut-S/GM-CSF while GM-CSF alone patients will be boosted with GM-CSF alone). Patient blinding will be maintained throughout the study.

Subjects will be followed for safety issues, immunologic response and clinical recurrence. Patients will be monitored 48-72 hours after each inoculation for reaction to the inoculation as well as documentation of any adverse effects experienced. Immunologic response will be monitored primarily by in vivo delayed type hypersensitivity (DTH) reactions but also may be documented by other immunologic assays. All patients will be followed for a total of 36 months from the time of initiation of trastuzumab maintenance therapy to document disease-free status.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1
* AJCC stage I - III non-inflammatory, HER2-positive (according to ASCO-CAP guidelines 5) breast cancer
* Completed neoadjuvant therapy with an approved regimen that includes trastuzumab and at least four cycles (12 weeks) of taxane-containing chemotherapy and underwent surgery with final pathology showing evidence of residual disease in the breast or axilla (residual ductal carcinoma in situ or microinvasive disease not eligible) or underwent surgery as a first intervention and was found to be pathologically node-positive: ≥ 4 positive lymph nodes (pN2 or pN3) regardless of hormone receptor status or 1-3 positive lymph nodes (pN1) if hormone receptor negative. Patients with micrometastases (pN1mi) are not eligible.
* Completed an approved regimen of neoadjuvant or adjuvant therapy with an approved regimen that includes trastuzumab and at least four cycles (12 weeks) of taxane-containing chemotherapy with plan for completion of one year of trastuzumab therapy.
* Completed appropriate surgical therapy to include:

  1. Total mastectomy and axillary staging with sentinel lymph node dissection or axillary lymph node dissection (level I/II). Patients with a positive sentinel lymph node must have undergone a completion axillary lymph node dissection.
  2. Breast conserving surgery (BCS) and axillary staging with sentinel lymph node dissection or axillary lymph node dissection. Patients undergoing surgery as a first intervention with a positive sentinel lymph node must have undergone a completion axillary dissection level I/II unless they had clinically node negative T1-T2 tumors and fewer than 3 involved lymph nodes. Patients receiving neoadjuvant chemotherapy that have a positive sentinel lymph node must have undergone a completion axillary lymph node dissection.
  3. Completed or receiving appropriate radiation therapy if indicated:

For patients undergoing total mastectomy surgery as a first intervention, post-mastectomy radiation to the chest wall, infraclavicular and supraclavicular areas is required for patients with ≥ 4 positive lymph nodes. Radiation to the internal mammary lymph nodes is not required per protocol but is allowed at the discretion of the patient's treating radiation oncologist. For patients with 1-3 positive lymph nodes, post-mastectomy radiation to the chest wall, infraclavicular, supraclavicular, and internal mammary areas is not required per protocol but is allowed at the discretion of the patient's treating radiation oncologist.

* For patients undergoing breast conserving surgery (BCS) as a first intervention, whole breast irradiation with or without a boost, and radiation to the infraclavicular and supraclavicular areas is required for patients with ≥ 4 positive lymph nodes. Radiation to the internal mammary lymph nodes is not required but is allowed at the discretion of the patient's treating radiation oncologist. For patients with 1-3 positive lymph nodes, whole breast irradiation with or without a boost is required. Radiation to the infraclavicular, supraclavicular, and internal mammary areas is not required per protocol but is allowed at the discretion of the patient's treating medical oncologist.
* For patient's undergoing mastectomy after neoadjuvant chemotherapy post-mastectomy radiation to the chest wall, infraclavicular and supraclavicular areas is required for patients presenting with clinical N2 or N3 disease or with ≥ 4 positive lymph nodes identified pathologically at the time of surgery. Radiation to the internal mammary lymph nodes is not required per protocol but is allowed at the discretion of the patient's treating radiation oncologist. For patients with 0-3 positive lymph nodes identified pathologically, post-mastectomy radiation to the chest wall, infraclavicular, supraclavicular and internal mammary areas is not required per protocol but is allowed at the discretion of the patient's treating radiation oncologist.
* For patient's undergoing BCS after neoadjuvant chemotherapy, whole breast irradiation with or without a boost is required. For patients with clinical N2 or N3 disease or with ≥ 4 positive lymph nodes identified pathologically at the time of surgery, radiation to the infraclavicular and supraclavicular areas is required. Radiation to the internal mammary lymph nodes is not required per protocol but is allowed at the discretion of the patient's treating radiation oncologist. For patients with 0-3 positive lymph nodes identified pathologically, radiation to the infraclavicular, supraclavicular and internal mammary areas is not required per protocol but is allowed at the discretion of the patient's treating radiation oncologist.

  * HLA-A2+ or HLA-A3+ or HLA-A24+ or HLA-A26+
  * LVEF >50%, or an LVEF within the normal limits of the institution's specific testing (MUGA or ECHO)
  * Adequate organ function as determined by the following laboratory values:

    1. ANC ≥ 1,000/μL
    2. Platelets ≥ 75,000/μL
    3. Hgb ≥ 9 g/dL
    4. Creatinine ≤ 1.5 x upper limit of normal (ULN) of institution's range or Creatinine clearance ≥ 50%
    5. Total bilirubin ≤ 1.5 ULN of institution's range
    6. ALT and AST ≤ 1.5 ULN of institution's range
    7. For women of child-bearing potential, agreement to use adequate birth control (abstinence, hysterectomy, bilateral oophorectomy, bilateral tubal ligation, oral contraception, IUD, or use of condoms or diaphragms)
  * Signed informed consent

Exclusion criteria:

* AJCC Stage IV breast cancer
* NYHA stage 3 or 4 congestive heart failure
* Immune deficiency disease or known history of HIV, HBV, HCV
* Receiving immunosuppressive therapy including chronic steroids, methotrexate, or other known immunosuppressive agents
* Pregnancy (assessed by urine HCG)
* Breast feeding
* Any active autoimmune disease requiring treatment, with the exception of vitiligo
* Active pulmonary disease requiring medication to include multiple inhalers (>3 inhalers including one containing steroids)
* Involved in other experimental protocols except with permission of other PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COL (ret) George E Peoples, MD, FACS, Study Director — LumaBridge
Locations (24):
- United States (24):
  - Sarcoma Oncology Research Center, LLC, Santa Monica, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Miami, Deerfield Beach, Florida
  - Memorial Breast Cancer Center, Hollywood, Florida
  - University of Miami, Kendall, Florida
  - University of Miami, Miami, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - University of Miami, Plantation, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Medstar Health (Union Memorial Hospital), Baltimore, Maryland
  - Medstar (Good Samaritan Hospital), Baltimore, Maryland
  - The Valley Hospital, Paramus, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Alliance/Presbyterian Cancer Center, Albuquerque, New Mexico
  - Tisch Cancer Institute/Icahn School of Medicine at Mount Sinai, New York, New York
  - North Shore Hematology Oncology Associates, The Bronx, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology (Cancer Care Centers of South Texas), San Antonio, Texas
  - University of Virginia Human Immune Therapy Center, Charlottesville, Virginia
  - Providence Regional Medical Center, Everett, Washington
  - Ascension/ Columbia St. Mary's, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab + NeuVax: Patients randomized to this arm will receive vaccinations of nelipepimut-S (1000 μg) and GM-CSF (250 μg) (NeuVax vaccine) administered intradermally every three weeks for six total vaccinations,
Period: Overall Study
Arm/Group | Trastuzumab + NeuVax | Trastuzumab + GM-CSF
Started | 50 | 50
Completed | 31 | 36
Not Completed | 19 | 14

BASELINE CHARACTERISTICS:
Groups:
- Trastuzumab + NeuVax: Patients randomized to this arm will receive vaccinations of nelipepimut-S (1000 μg) and GM-CSF (250 μg) (NeuVax vaccine) administered intradermally every three weeks for six total vaccinations,
  Trastuzumab: Herceptin will be administered to patients every three weeks as monotherapy for one year,
  GM-CSF: For patients randomized to the GM-CSF alone arm, they will receive inoculations of GM-CSF (250mcg) administered intradermally every three weeks for six total vaccinations,
- Trastuzumab + GM-CSF: Patients randomized to this arm will receive inoculations of GM-CSF (250 μg) administered in an identical manner to those receiving nelipepimut-S/GM-CSF (NeuVax). Patients will be blinded as to whether they are receiving nelipepimut-S/GM-CSF or GM-CSF alone.
  Trastuzumab: Herceptin will be administered to patients every three weeks as monotherapy for one year, to be given upon completion of standard of care chemotherapy/radiotherapy.
  GM-CSF: For patients randomized to the GM-CSF alone arm, they will receive inoculations of GM-CSF (250mcg) administered intradermally every three weeks for six total vaccinations,
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + NeuVax | Trastuzumab + GM-CSF | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 44 | 86
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 7 | 10
  White | 33 | 29 | 62
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-free Survival (DFS)
Description: Compare invasive DFS between the two treatment groups from time of initiation of trastuzumab maintenance therapy (trasuzumab monotherapy) to time of invasive local, regional or distant recurrence, new primary, or death due to any cause. Disease state will be determined by the patients' own physicians at the individual study sites during their routine follow-up screening. This will occur for all enrolled patients, regardless of randomization, approximately every three months for the first 24 months after completion of primary therapies and every six months thereafter with clinical exam, and laboratory and radiographic surveillance. The primary outcome measure of the trial is invasive DFS.
Time Frame: Initiation of trastuzumab monotherapy through the end of the patient's fifth year of participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab + NeuVax | Trastuzumab + GM-CSF
Number analyzed (Participants) | 50 | 50
Participants | 42 | 47

2. Secondary Outcome: Local and Systemic Toxicities
Description: Standard local and systemic toxicities will be collected and graded per the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 graded toxicity scale. For both the inoculations during the primary vaccine/inoculation series and the booster inoculations, patients will be monitored closely for one hour after inoculation with questioning, serial exams and vital signs every 15 minutes to observe for a hypersensitivity reaction. Additionally, patients will return to their study site 48-72 hours after inoculation for questioning regarding any systemic toxicity and local injection site reactions. When they return to their study site, the local reaction at the inoculation sites will be examined and measured.
Time Frame: From the date of initiation of the vaccine or inoculation series and booster series up to 36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab + NeuVax | Trastuzumab + GM-CSF
Number analyzed (Participants) | 50 | 50
Participants | 46 | 43

3. Secondary Outcome: Evaluate in Vivo and in Vitro Immune Responses
Description: Immune responses will be primarily documented using the delayed type hypersensitivity (DTH) reaction and using the dextramer assay to enumerate peptide-specific CTL. Each of these measurements will be performed regardless of randomization. DTH reactions will be measured prior to initiation of the primary vaccine/inoculation series, one month ± 1 week after completion of the primary vaccine/inoculation series, and one month ± 1 week after the final booster inoculation. Dextramer measurements will be performed prior to initiating the primary vaccine/inoculation series as well as one month ± 1 week after completion of the vaccine/inoculation series. Additionally, these assays may be performed pre- and post-each booster. Alternatively, these assayed time points may also be performed all at once on frozen and banked cells.
Time Frame: From the date of the first inoculation of Trastuzumab monotherapy to the end of the patient's fifth year of participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab + NeuVax | Trastuzumab + GM-CSF
Number analyzed (Participants) | 50 | 50
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Trastuzumab + NeuVax | Trastuzumab + GM-CSF
All-Cause Mortality (participants affected / at risk) | 0/50 | 1/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 5/50
Other Adverse Events (participants affected / at risk) | 43/50 | 38/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab + NeuVax (N=50) | Trastuzumab + GM-CSF (N=50)
Left Breast Infection (Infections and infestations) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Procedural Complication-Tram Flap Failure (Surgical and medical procedures) | 0 (0) | 1 (1)
Sepsis (General disorders) | 1 (1) | 0 (0)
UTI - Pyelonephritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab + NeuVax (N=50) | Trastuzumab + GM-CSF (N=50)
Pruritus (Infections and infestations) | 6 (6) | 4 (4)
Injection site reaction-Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
Headache (Nervous system disorders) | 6 (6) | 3 (3)
Fatigue (General disorders) | 3 (3) | 5 (5)
Pain Injection Site (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Fever (General disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Withdrawls (General disorders) | 7 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02297698/Prot_SAP_000.pdf